CLINICAL TRIAL: NCT05351749
Title: Implementing Prescriber-Pharmacist Collaborative Care for Evidence-based Anticoagulant Use
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Geoffrey Barnes, Assistant Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: HUM00207165; R18HS028562 (AHRQ)
Record Dates: First submitted 2022-04-06; First posted 2022-04-28 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Embolism; Venous Thromboembolism; Atrial Fibrillation
Keywords: Prescribing alerts; Anticoagulation
MeSH Terms: conditions — Pulmonary Embolism; Venous Thromboembolism; Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- New-prescription Alert / Existing-prescription notification to prescriber (Experimental)
  Interventions: Behavioral: New-prescription Alert; Behavioral: Existing-prescription notification to prescriber
- New-prescription Alert w/ referral option/ Existing-prescription notification to prescriber (Experimental)
  Interventions: Behavioral: New-prescription Alert with referral option; Behavioral: Existing-prescription notification to prescriber
- New-prescription Alert/ Existing-prescription notification to pharmacist (Experimental)
  Interventions: Behavioral: New-prescription Alert; Behavioral: Existing-prescription notification to pharmacist
- New-prescription Alert w/ referral option/ Existing-prescription notification to pharmacist (Experimental)
  Interventions: Behavioral: New-prescription Alert with referral option; Behavioral: Existing-prescription notification to pharmacist

INTERVENTIONS:
Behavioral: New-prescription Alert — An enhanced drug alert notification in the Michigan Medicine electronic health record (EHR) that is tailored to the specific type of inappropriate Direct Oral Anticoagulant (DOAC) use (e.g., dosing too high for renal dysfunction) and offers decision support to the prescriber to alter a newly prescribed DOAC prescription.
  Arms: New-prescription Alert / Existing-prescription notification to prescriber; New-prescription Alert/ Existing-prescription notification to pharmacist
Behavioral: New-prescription Alert with referral option — An enhanced drug alert notification in the EHR that is tailored to the specific type of inappropriate DOAC use (e.g., dosing too high for renal dysfunction) and offers decision support to the prescriber to alter new DOAC prescription. This alert will ALSO include an option for referral to the anticoagulation clinic pharmacist for assistance.
  Arms: New-prescription Alert w/ referral option/ Existing-prescription notification to pharmacist; New-prescription Alert w/ referral option/ Existing-prescription notification to prescriber
Behavioral: Existing-prescription notification to prescriber — Prescriber receives a notification through the EHR indicating an existing DOAC prescription may not be appropriate (e.g. due to renal function change, new drug-drug interactions), and recommending a prescription update.
  Arms: New-prescription Alert / Existing-prescription notification to prescriber; New-prescription Alert w/ referral option/ Existing-prescription notification to prescriber
Behavioral: Existing-prescription notification to pharmacist — Pharmacist receives a notification through the EHR indicating an existing DOAC prescription may not be appropriate (e.g. due to renal function change, new drug-drug interactions), and recommending a prescription update.
  Arms: New-prescription Alert w/ referral option/ Existing-prescription notification to pharmacist; New-prescription Alert/ Existing-prescription notification to pharmacist

SUMMARY:
The researchers hypothesize that existing-prescription notifications directed to pharmacists are more likely to lead to a prescription change than existing-prescription notifications directed to prescribers. Furthermore, the researchers hypothesize that the availability of a pharmacist referral option is associated with a higher rate of prescription changes for initial-prescription alerts that are directed to the prescriber at the time of initial-prescribing errors.

Findings from this project will establish a framework for implementing prescriber-pharmacist collaboration for high risk medications, including anticoagulants

DETAILED DESCRIPTION:
Please note that the 3rd and 4th outcome measures are conditional on the outcomes of the 1st and 2nd outcome measures respectively.

Please note that enrollment of 300 will provide sufficient power to study.

ELIGIBILITY:
Prescribers:

Inclusion Criteria:

* Michigan Medicine provider with prescribing privileges
* Providers in ambulatory care settings
* Prescribe DOAC to patients 18 years and older

Exclusion Criteria:

* Providers in inpatient settings
* Providers who are members of the study team

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
The number (proportion) of notifications (in the existing-prescription notification conditions) that are addressed within 7 days. | Up to 7 days
  Existing-prescription notification conditions = Prescriber notification & Pharmacist notification

SECONDARY OUTCOMES:
The number (proportion) of alerts (in the newly prescribed DOAC alert conditions) that are addressed within 7 days. | Up to 7 days
  Newly prescribed DOAC alert conditions= Medication alert & Medication alert + referral
Change in effect size for the existing-prescription notification over time | Month 0, Up to 18 months
  Reported on at the institution level (not individual level). Existing-prescription notification conditions = Prescriber notification & Pharmacist notification
  This outcome measure analysis is based on the results of outcome #1.
Change in effect size for the initial alert over time | Month 0, Up to 18 months
  Reported on at the institution level (not individual level). Newly prescribed DOAC alert condition= Medication alert & Medication alert + referral
  This outcome measure analysis is based on the results of outcome #2.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Barnes, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barnes GD, Choi SY, Lanham MS, Dorsch MP, Errickson J, Fabbri M, Saraswat A, Seagull FJ, Smith SN. Implementing prescriber-pharmacist collaboration to improve evidence-based medication prescribing using asynchronous, non-interruptive electronic health record notifications. Implement Sci. 2025 Dec 15. doi: 10.1186/s13012-025-01478-9. Online ahead of print. PMID 41398697
- [Derived] Smith SN, Lanham MSM, Seagull FJ, Fabbri M, Dorsch MP, Jennings K, Barnes G. System-Wide, Electronic Health Record-Based Medication Alerts for Appropriate Prescribing of Direct Oral Anticoagulants: Pilot Randomized Controlled Trial. JMIR Form Res. 2024 Nov 8;8:e64674. doi: 10.2196/64674. PMID 39514247
- [Derived] Smith SN, Lanham M, Seagull FJ, Dorsch M, Errickson J, Barnes GD. Implementing pharmacist-prescriber collaboration to improve evidence-based anticoagulant use: a randomized trial. Implement Sci. 2023 May 15;18(1):16. doi: 10.1186/s13012-023-01273-4. PMID 37189171